CLINICAL TRIAL: NCT05113771
Title: A Biomarker-Guided, Randomized, Double-Blind, Placebo-Controlled Efficacy and Safety Study of Liafensine in Patients With Treatment-Resistant Depression
Brief Title: A Biomarker-Guided, Randomized, Placebo-Controlled Efficacy and Safety Study of Liafensine in Patients With TRD
Acronym: ENLIGHTEN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Denovo Biopharma LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DB104-01
Record Dates: First submitted 2021-10-29; First posted 2021-11-09 (Actual); Results first posted 2025-05-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-03

CONDITIONS: Treatment Resistant Depression
Keywords: TRD, Treatment Resistant Depression
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Liafensine 1mg (Experimental): Patients with TRD were treated with liafensine 1 mg QD for 6 weeks.
  Interventions: Drug: Liafensine
- Liafensine 2mg (Experimental): Patients with TRD were treated with liafensine 2 mg QD for 6 weeks.
  Interventions: Drug: Liafensine
- Placebo (Placebo Comparator): Patients with TRD were treated with placebo 1 mg QD for 6 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Liafensine — Liafensine
  Other Names: DB104
  Arms: Liafensine 1mg; Liafensine 2mg
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This study was conducted as a randomized, double-blind, placebo-controlled, multi-center Phase 2b study. Approximately 180 subjects with treatment resistant depression who meet all eligibility criteria will be enrolled. The primary endpoint is to demonstrate liafensine is superior to placebo in DGM4 positive patients with TRD.

DETAILED DESCRIPTION:
This study is a randomized, double blind, placebo-controlled Phase 2b study to assess the efficacy, safety, tolerability, and pharmacokinetics of liafensine. Eligible patients were randomized 1:1:1 to receive liafensine 1 mg QD, liafensine 2 mg QD, or placebo QD. The main objectives of this study are as follows:

Primary Efficacy Objective: To demonstrate that liafensine was superior to placebo in DGM4 positive patients with TRD as assessed by the change in MADRS total score from baseline to Day 42 of double blind treatment

Key Secondary Efficacy Objective: To evaluate the change from baseline to Day 42 in DGM4 positive patients with TRD treated with liafensine vs placebo on the Clinical Global Impression-Severity Scale (CGI S)

Other Secondary Efficacy Objective: To evaluate the Clinical Global Impression-Improvement Scale (CGI I) at Day 42 in DGM4 positive patients with TRD treated with liafensine vs placebo

Safety Objective: To compare the safety and tolerability of liafensine vs placebo in all randomized patients with TRD who received at least one dose of study drug during double blind treatment

Psychiatric assessments were performed by a psychiatrist or trained and certified clinical staff member. Neurologic assessments were performed by an experienced clinician. Patients who fulfilled Hy's Law, defined as ALT or AST ≥ 3 × ULN and TBL ≥ 2 × ULN, in the absence of significant increase in ALP and in the absence of an alternative diagnosis that explained the increase in total bilirubin, were discontinued, with medical follow up as appropriate.

ELIGIBILITY:
Inclusion Criteria:

1. Provide signed informed consent which includes pharmacogenomic (PGx) testing.
2. Have a diagnosis of MDD without psychotic features, according to the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) criteria, based on clinical assessment and confirmed by the Mini International Neuropsychiatric Interview (MINI).
3. Have a history of TRD within the past 5 years as documented by the Massachusetts General Hospital (MGH) Antidepressant Treatment Response Questionnaire (ATRQ) (5-year version). That is, within the past 5 years study participants must have had a clinically meaningful inadequate response (estimated < 50% improvement per Investigator/patient consensus and documented by the Investigator) to at least two treatment courses with antidepressant regimens. These must involve at least two different pharmacologic treatment classes* and have been given at accepted therapeutic doses for an adequate duration (at least 6 weeks). One of these treatment failures must have occurred within the current episode.

   *Note: Non-pharmacological treatment (eg, cognitive behavioral therapy, electroconvulsive therapy, repetitive transcranial magnetic stimulation, vagus nerve stimulation, acupuncture) are not counted as treatment regimen.
4. To be eligible, patients must have DGM4 genotype results obtained from the designated Clinical Laboratory Improvement Amendments (CLIA) lab, and all eligible DGM4-positive patients and about 20% DGM4-negative patients will be randomly included by an IRT system in order to achieve the appropriate randomization ratio of DGM4-positive vs negative patients.
5. Pregnancy conception limitations

   * Female patients must be postmenopausal or surgically sterile or, if of childbearing potential and the partner is not vasectomized (6 months minimum), must agree to use a medically acceptable form of contraception from the time of signing the informed consent form (ICF) through at least 60 days following the last administration of study drug. If only the barrier method is used, a double barrier must be employed. Postmenopausal women must have had ≥ 24 months of spontaneous amenorrhea. Surgically sterile women are defined as those who have had a hysterectomy, bilateral ovariectomy, or bilateral tubal ligation. All women of childbearing potential must have a negative pregnancy test result before administration of study drug.
   * Male patients must be biologically incapable of having children (eg, vasectomized) or must agree to use the above forms of birth control for themselves and their partner from the time of signing the informed consent form through at least 120 days following the last administration of study drug.
6. Be fluent in the local language.
7. Male or female aged 18 to 70, inclusive, at time of enrollment.
8. Have a HAMD-17 total score ≥ 21 at screening.
9. Be willing to discontinue the use of antidepressant drugs (including over-the-counter medications to treat depression [eg, St John's Wort]) at least 5 half-lives (or at least 1 week for herbal or other over-the-counter medications for depression) prior to baseline (Day -1). For fluoxetine, a washout period of at least 3 weeks for ≤ 20 mg/day and at least 4 weeks for > 20 mg/day is required.

Exclusion Criteria:

1. Prior participation in a study with liafensine
2. Used any investigational drug product, device, or biologic within 6 months or five half-lives (whichever is longer) prior to baseline (Day -1).
3. A positive pregnancy test result or currently breastfeeding.
4. Clinically significant illness (including chronic, persistent, or acute infection), medical/surgical procedure, or trauma within 30 days prior to screening or between screening and baseline (Day 1) as determined by the investigator.
5. A history or presence of a clinically significant hepatic, renal, gastrointestinal, cardiovascular, endocrine, respiratory, immunologic, hematologic, dermatologic, or neurologic abnormality, or any other condition, that in the investigator's opinion, represent potential risk to the patient's safety, full participation in the study, or affect the absorption, distribution, metabolism, or excretion of liafensine.
6. Presence of autoimmune hepatitis, primary sclerosing cholangitis, untreated hepatitis C, active hepatitis B, or any other uncontrolled or unstable liver disease according to local guidance.
7. Uncontrolled human immunodeficiency virus (HIV) infection according to local guidance.
8. Uncontrolled abnormal thyroid function according to local guidance.
9. One or more clinical laboratory evaluations are outside the reference range, at screening, that are in the investigator's opinion, of potential risk to the patient's safety.
10. Has at the Screening Visit:

    * Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) levels > 1.5x the upper limit of normal (ULN) at screening.
    * Total bilirubin (TBL) > 2 mg/dL (34.2 μmol/L) at screening, unless there is an explained indirect hyperbilirubinemia, eg, Gilbert's syndrome.
    * Alkaline phosphatase (ALP) > 1.5x the ULN at screening. Note: Laboratory tests can be repeated to see if values return to normal range, but any such laboratory abnormality must be resolved by the Baseline Visit (Day -1).
11. Clinically significant vital sign abnormality at screening. This includes, but is not limited to, the following, in the supine (after at least 5 min rest) and standing (after 1 min and 3 min standing): systolic blood pressure ≥ 140 mmHg; diastolic blood pressure ≥ 90 mmHg; or heart rate < 50 or > 90 beats per minute. If the initial blood pressure is ≥ 140/90 mmHg, the lowest value from up to 3 additional attempts, which also must not be ≥ 140/90 mmHg, should be used. Patients with symptomatic orthostatic hypotension, at the discretion of investigator, will be excluded.
12. Corrected QT interval measurement according to the Fridericia rule (QTcF) > 450 msec for men and > 470 msec for women during controlled rest at screening, or history of long-QT syndrome.
13. ECGs containing any of the following readings:

    * Left bundle branch block
    * Right bundle branch block with QRS duration > 140 ms
    * Intraventricular conduction defect with QRS duration > 140 ms
    * Long QT syndrome
14. History of seizure, other than childhood febrile seizures.
15. History of clinically significant head trauma, including closed head injury with loss of consciousness, that is, in the opinion of the investigator, likely to affect central nervous system function.
16. History of clinically significant symptomatic orthostatic hypotension (ie, postural syncope).
17. History of narrow angle glaucoma.
18. History of cancer within 2 years prior to screening or between screening and baseline (Day -1), except for non-metastatic basal and/or squamous cell carcinoma of the skin.
19. Use of prescription or nonprescription medications for attention-deficit hyperactivity disorder (ADHD), narcolepsy, or cognitive enhancement (eg, methylphenidate, atomoxetine, modafinil, ginkgo biloba, and huperzine A) within 30 days prior to screening or between screening and baseline (Day -1).
20. Regular consumption of (eg, more days than not) excessive quantities of xanthine-containing beverages (eg, more than five cups of coffee or the equivalent per day) within 30 days prior to screening or between screening and baseline (Day -1).
21. Urine drug screen (UDS) positive for a drug of abuse, with the exception of cannabis in countries where it is legally available (see Table 3 for list of drugs of abuse). Where legal, prior use of cannabis is permitted provided the patient agrees to abstain from smoking or ingesting cannabis or cannabis products during the study.
22. Use of potent inducers of CYP3A4 (eg, rifampin, rifabutin, phenytoin, carbamazepine, or phenobarbital) within 2 weeks prior to baseline (Day-1).
23. Current diagnosis or history of a psychotic disorder, MDD with psychotic features, manic or hypomanic episode of bipolar or related disorders.
24. Current diagnosis of anxiety disorder (if primary), post-traumatic stress disorder, obsessive compulsive disorder (if primary), intellectual disability (DSM-5 diagnostic code 319), borderline personality disorder, antisocial personality disorder, histrionic personality disorder, or narcissistic personality disorder according to the DSM-5 criteria, or any other psychiatric or neurologic disorder or symptom due to a general medical condition, that, in the judgement of the investigator, could pose undue risk to the patient or compromise the study.
25. Hospitalized or discharged from psychiatric ward within 8 weeks prior to the screening visit and planned hospitalization for any condition(s) during the study.
26. Moderate or severe alcohol use disorder or other substance use disorder (except nicotine or caffeine), within 6 months prior to screening, according to the DSM-5 criteria.
27. Significant risk of suicide determined by:

    1. Acute suicidality as evidenced by answering "yes" to Question 5 ("In the Past Year") on the C-SSRS, indicating active suicidal ideation with specific plan and intent for suicide, at screening, or baseline (Day -1); or
    2. History of suicidal behavior as indicated by a "yes" response on the Suicidal Behavior section of the C-SSRS ("In the past year") or
    3. A score ≥ 5 on Item 10 (suicidal thoughts) of the MADRS at screening or baseline (Day -1); or
    4. Has attempted suicide within 6 months prior to the initial screening visit.
28. Previous allogenic bone marrow transplant.
29. Received non-leukocyte-depleted whole blood transfusion within 4 months prior to PGx testing at Screening.
30. Currently employed by the sponsor or by a clinical trial site participating in this study, or a first-degree relative of an employee of the sponsor or of an employee at a participating clinical trial site.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2022-06-29 (Actual); Primary Completion 2024-02-06 (Actual); Study Completion 2024-03-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew A Spear, M.D., Study Director — Denovo Biopharma
Locations (44):
- United States (40):
  - University of Alabama at Birmingham, Huntsville, Alabama
  - Alea Research, Phoenix, Arizona
  - Collaborative Neuroschience Research, LLC, Garden Grove, California
  - Behavioral Research Specialists, LLC, Glendale, California
  - Sunwise Clinical Research, LLC., Lafayette, California
  - Excell Research, Oceanside, California
  - Anderson Clinical Reseach, Redlands, California
  - Schuster Medical Research Institute, Sherman Oaks, California
  - Collaborative Neuroscience Research, LLC, Torrance, California
  - Pacific Clinical Research Management Group, Upland, California
  - Clinical Research of Brandon, LLC, Brandon, Florida
  - Access Research Institute, Brooksville, Florida
  - The Medicine Medical Research, Hollywood, Florida
  - Nuovida Research Center, Miami, Florida
  - SG Research, LLC, Miami, Florida
  - Aqualane Clinical Research, Naples, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - CenExel Atlanta Center for Medical Research, Atlanta, Georgia
  - Psych Atlanta, PC, Marietta, Georgia
  - Revive Research Institute, Inc, Elgin, Illinois
  - Ascension Via Christi Research, a division of Ascension Via Christi Hospitals Wichita, Inc., Wichita, Kansas
  - Pharmasite Research, Inc., Baltimore, Maryland
  - CBH Health LLC, Gaithersburg, Maryland
  - Boston Clinical Trials & Medical Research, Boston, Massachusetts
  - Neurobehavioral Medicine Group, Bloomfield, Michigan
  - Alivation Research, LLC, Lincoln, Nebraska
  - Altea Research Institute, Las Vegas, Las Vegas, Nevada
  - Hassman Research Institute, Marlton, New Jersey
  - Global Medical Institutes, LLC, Princeton, New Jersey
  - Bio Behavior Health, Toms River, New Jersey
  - IMA Clinical Research, Albuquerque, New Mexico
  - Zucker Hillside Hospital, Glen Oaks, New York
  - The Ohio State University Department of Psychiatry, Columbus, Ohio
  - Lehigh Center for Clinical Research, LLC, Allentown, Pennsylvania
  - Global Medical Institutes, LLC, Moosic, Pennsylvania
  - FutureSearch Trials of Dallas, Dallas, Texas
  - InSite Clinical Research, DeSoto, Texas
  - North Texas Clinical Trials, Fort Worth, Texas
  - University of Texas Medical School at Houston, Houston, Texas
  - Core Clinical Research, Everett, Washington
- Canada (4):
  - OCT Research ULC, Kelowna, British Columbia
  - AMNDX Inc., Markham, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - CAMH-Russell Street Site 250 College Street, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang G, Aguado M, Spear MA, Alphs L, Chen C, Huang H, Lu XX, Doostzadeh J, Wu S, Wang S, Patel A, Nemeroff CB, Wang Z, Li A, Luo W. ANK3 as a Novel Genetic Biomarker for Liafensine in Treatment-Resistant Depression: The ENLIGHTEN Randomized Clinical Trial. JAMA Psychiatry. 2025 Dec 1;82(12):1186-1194. doi: 10.1001/jamapsychiatry.2025.2416. PMID 40928787

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Intent to treat (ITT) population 196 (65 participants in Liafensine 1mg arm, 64 patients in Liafensine 2mg arm, and 67 patients in placebo arm). Total 197 patients were initially randomized, but one patient was not dosed.
Period: Overall Study
Arm/Group | Liafensine 1mg | Liafensine 2mg | Placebo
Started | 65 | 65 | 67
Intent To Treat (ITT): All Patients Who Took at Least One Dose | 65 | 64 | 67
DGM4Positive Analysis Set: Patients Who Took at Least 1 Dose Study Drug & Had an Efficacy Evaluation | 62 | 61 | 63
Completed | 61 | 49 | 52
Not Completed | 4 | 16 | 15

BASELINE CHARACTERISTICS:
Population: Intent to treat (ITT) population is equal to196 (65 participants in liafensine 1mg arm, 64 patients in liafensine 2mg arm, and 67 patients in placebo arm), which is including all patients who took at least 1 dose of study drug. Total of 197 patients were initially randomized and one randomized patient was not dosed.
Groups:
- Total: Total of all reporting groups
Arm/Group | Liafensine 1mg | Liafensine 2mg | Placebo | Total
Number analyzed (Participants) | 65 | 64 | 67 | 196
Age, Categorical [Count of Participants; unit: Participants] — Population: Intent to treat (ITT) population is equal to196 (65 participants in liafensine 1mg arm, 64 patients in liafensine 2mg arm, and 67 patients in placebo arm), which is including all patients who took at least 1 dose of study drug. Total of 197 patients were initially randomized and one randomized patient was not dosed.
  Participants
    <=18 years | 0 | 0 | 0 | 0
    Between 18 and 65 years | 55 | 60 | 62 | 177
    >=65 years | 10 | 4 | 5 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Intent to treat (ITT) population is equal to196 (65 participants in liafensine 1mg arm, 64 patients in liafensine 2mg arm, and 67 patients in placebo arm), which is including all patients who took at least 1 dose of study drug. Total of 197 patients were initially randomized and one randomized patient was not dosed.
  years | 43.6 (15.47) | 42.2 (13.96) | 43.9 (14.81) | 43.2 (14.71)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Intent to treat (ITT) population is equal to196 (65 participants in liafensine 1mg arm, 64 patients in liafensine 2mg arm, and 67 patients in placebo arm), which is including all patients who took at least 1 dose of study drug. Total of 197 patients were initially randomized and one randomized patient was not dosed.
  Participants
    Female | 41 | 45 | 36 | 122
    Male | 24 | 19 | 31 | 74
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Intent to treat (ITT) population is equal to196 (65 participants in liafensine 1mg arm, 64 patients in liafensine 2mg arm, and 67 patients in placebo arm), which is including all patients who took at least 1 dose of study drug. Total of 197 patients were initially randomized and one randomized patient was not dosed.
  Participants
    Asian | 33 | 32 | 32 | 97
    Black or African American | 1 | 0 | 2 | 3
    white | 31 | 32 | 32 | 95
    other | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 30 | 33 | 32 | 95
  Canada | 3 | 0 | 3 | 6
  China | 32 | 31 | 32 | 95

OUTCOME MEASURES:

1. Primary Outcome: Change in Montgomery Åsberg Depression Rating Scale (MADRS) Total Score From Baseline to Day 42, in DGM4-positive Patients
Description: The primary objective of this study was change of Montgomery Åsberg Depression Rating Scale (MADRS) total score (range = 0 60, with higher scores indicating more severe depression) in DGM4 positive patients who were treated with liafensine versus placebo.
Time Frame: Baseline to Day 42
Measure: Mean (Standard Error); unit: Units on a Scale
Groups:
- Liafensine 1mg or 2 mg: Patients with TRD were treated with liafensine 1 mg or 2mg QD for 6 weeks.
  Treatment: Liafensine
Arm/Group | Liafensine 1mg | Liafensine 2mg | Liafensine 1mg or 2 mg | Placebo
Number analyzed (Participants) | 62 | 61 | 123 | 63
Units on a Scale | -15.4 (1.25) | -15.5 (1.30) | -15.4 (0.90) | -11.0 (1.31)
Statistical Analysis 1: Comparison: Liafensine 1mg or 2 mg vs Placebo; Test type: Superiority; p = 0.0056, MMRM; mixed model for repeated measures (MMRM) with imputation based on the missing at random (MAR) assumption was used; LS Mean Difference = -4.4, 95% CI 2-sided [-7.6 to -1.3]

2. Secondary Outcome: Change From Baseline to Day 42 in Clinical Global Impression-Severity Scale (CGI-S) Score in DGM4 Positive Patients
Description: The secondary endpoint was the change from baseline to Day 42 in Clinical Global Impression-Severity Scale CGI-S score (range = 1-7, with higher scores indicating greater illness) in DGM4 positive patients.
Time Frame: Baseline to Day 42
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Groups:
- Liafensine 1mg or 2mg: Patients with TRD were treated with liafensine 1 mg or 2mg QD for 6 weeks.
  Treatment: Liafensine
Arm/Group | Liafensine 1mg | Liafensine 2mg | Liafensine 1mg or 2mg | Placebo
Number analyzed (Participants) | 62 | 61 | 123 | 63
Units on a scale | -1.5 (0.15) | -1.5 (0.16) | -1.5 (0.11) | -1.1 (0.15)
Statistical Analysis 1: Comparison: Liafensine 1mg or 2mg vs Placebo; Test type: Superiority; p = 0.0189, MMRM

3. Secondary Outcome: The Clinical Global Impression-Improvement Scale (CGI-I) (Range = 1-7, With Higher Score Indicating Worsening) Was Assessed in DGM4 Positive Patients
Description: To evaluate the Clinical Global Impression-Improvement Scale (CGI I) (range = 1-7, with higher score indicating worsening) at Day 42 in DGM4 positive patients with TRD treated with liafensine vs placebo
Time Frame: 42 days
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Liafensine 1mg and 2mg: Patients with TRD were treated with liafensine 1 mg or 2mg QD for 6 weeks.
  Treatment: Liafensine
Arm/Group | Liafensine 1mg | Liafensine 2mg | Liafensine 1mg and 2mg | Placebo
Number analyzed (Participants) | 62 | 61 | 123 | 63
units on a scale | 2.3 (0.88) | 2.4 (1.08) | 2.3 (0.97) | 2.9 (1.28)
Statistical Analysis 1: Comparison: Liafensine 1mg and 2mg; Test type: Superiority; p = 0.0026, Cochran-Mantel-Haenszel

ADVERSE EVENTS:
Time Frame: 42 days
Description: Treatment Emergent Adverse Events (TEAEs) (Safety Analysis Set) was performed. One randomized patient was not dosed.
Arm/Group | Liafensine 1mg | Liafensine 2mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/65 | 1/64 | 0/67
Serious Adverse Events (participants affected / at risk) | 0/65 | 3/64 | 2/67
Other Adverse Events (participants affected / at risk) | 36/65 | 37/64 | 38/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Liafensine 1mg (N=65) | Liafensine 2mg (N=64) | Placebo (N=67)
Ankle Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Hip Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Rib Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0
Intestinal Haematoma (Vascular disorders) | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 2
Death (General disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liafensine 1mg (N=65) | Liafensine 2mg (N=64) | Placebo (N=67)
Headach (Nervous system disorders) | 20 (65) | 14 | 15
Somnolence (Nervous system disorders) | 5 | 6 | 1
Dizziness (Nervous system disorders) | 8 | 2 | 5
Nausea (Gastrointestinal disorders) | 11 | 5 | 7
Constipation (Gastrointestinal disorders) | 7 | 6 | 0
Abdominal distension (Gastrointestinal disorders) | 5 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 4 | 1 | 1
Anxiety (Psychiatric disorders) | 5 | 0 | 2
Depression (Psychiatric disorders) | 0 | 1 | 5
Upper respiratory tract infection (Infections and infestations) | 1 | 5 | 3
Influenza (Infections and infestations) | 4 | 1 | 1
Fatigue (General disorders) | 4 | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 4 | 6 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 3 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-08-29): https://cdn.clinicaltrials.gov/large-docs/71/NCT05113771/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-18): https://cdn.clinicaltrials.gov/large-docs/71/NCT05113771/SAP_001.pdf